CLINICAL TRIAL: NCT00292695
Title: A Phase II Study of Concurrent Chemoradiation for The Localized Nasal NK/T-cell Lymphoma
Brief Title: A Phase II Study of Nasal NK/T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Mackay Memorial Hospital (Other); National Cheng-Kung University Hospital (Other); Taichung Veterans General Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Kaohsiung Veterans General Hospital. (Other); National Taiwan University Hospital (Other); Tri-Service General Hospital (Other); Chi Mei Medical Hospital (Other); Kaohsiung Medical University (Other); Changhua Christian Hospital (Other); Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1405
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Etoposide; Cisplatin; Ifosfamide; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chemoradiation (Experimental): Chemoradiation: IF-RT 50.4 Gy/28 Fractions, DEP: (Q4W, CCRT) X 2 Dexamethosone 20 mg/m2/d iv D1-3 VP-16 (etoposide) 75 mg/m2 iv 1 hr D1-3 Cisplatin 75 mg/m2 ivd 4 hr D1
  Interventions: Other: VP-16, Cisplatin, Ifosfamide, Dexamethosone, Mesna, IF-RT

INTERVENTIONS:
Other: VP-16, Cisplatin, Ifosfamide, Dexamethosone, Mesna, IF-RT — IF-RT 50.4 Gy/28 Fractions, DEP: (Q4W, CCRT) X 2 Dexamethosone 20 mg/m2/d iv D1-3 VP-16 (etoposide) 75 mg/m2 iv 1 hr D1-3 Cisplatin 75 mg/m2 ivd 4 hr D1
  DVIP: (Q4W, POST-RT) X 2 Dexamethosone 20 mg/m2/d iv D1-4 VP-16 (etoposide) 75 mg/m2 iv 1 hr D1-4 Ifosfamide 1.2 gm/m2/d ivd 2 hr D1-4 Mesna 240 mg/m2/d iv at 0, 4, 8 hr D1-4 Cisplatin 20 mg/m2 ivd 1 hr D1-4 G-CSF 250ug subcut D 9-12

SUMMARY:
To determine whether adding combinational chemotherapy concurrently to conventional radiation will improve the response rate, event-free survival, and overall survival.

To test the dose intensity and toxicity of chemotherapy in concurrence with radiation.

To detect the blood EBV DNA level in Chinese Nasal NK/T-cell lymphoma patients and correlate to the treatment response and prognosis.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Histologically proven extranodal NK/T-cell lymphoma, nasal type according to the WHO classification (must be pathology-proven EBV DNA positive as well as cytoplasmic CD3 +, while CD56+ is not an essential diagnostic criteria. ). Both newly diagnosed patients and who were previous chemotherapy-treated patients with residual or recurrent diseases will be allowed.
2. Any of lymphomatous involvement exist in nasal cavity and/or paranasal sinuses, orbit, Waldeyer's ring, and oral cavity PS with ECOG scale 0-2.
3. Stage I or contiguous stage II, measurable or evaluable lymphoma by clinical imaging No previous chemotherapy and/or radiotherapy.
4. ANC ≧ 2,000/mm3, Platelet ≧ 100,000/mm3 of peripheral blood.
5. Age <70.
6. Total bilirubin < 2.5 mg/dl Serum creatinine ≦1.5 mg/dl Blood urea nitrogen (BUN) ≦ 25 mg/dl
7. Signed informed consent

Exclusion criteria:

1. Pregnancy or lactation period
2. Severe intercurrent illness, e.g. infection, heart failure
3. Myocardial infarction within recent 12 months
4. Known hypersensitivity to any component drug of the treatment regimen

TREATMENT PLAN

Concurrent chemoradiation is the primary treatment. The treatment will be started within 2 weeks after registration. The patients are intended to receive the complete radiation dose (50 Gy) and 2 courses of DEP regimen concurrently. The first course of DEP regimen must be started within one week before or after the initiation of radiation (1st week). The second course of DEP regimen will be given in 4 weeks (i.e. the 5th week) after completion of the first course of DEP and during the period of radiotherapy. The first evaluation of response by CT or MRI will be performed at 4 weeks after the completion of the second course DEP (i.e. the 9th week). If patients respond to therapy or remain in the SD situation, DVIP regimen will be followed immediately every 4 weeks for another 2 courses as a consolidation therapy. If patients are progressive, study treatment will be stopped and patients will be off-studied. And they will proceed to salvage therapy with DHAP regimen for ethical reason. The second evaluation of response will be performed in 4 weeks after completion of treatment (i.e. 21st week).

1. Systemic chemotherapy with DEP and DVIP regimens

   Schedule and Dose for DEP (q4w, CCRT) Dexamethosone 20 mg/m2/d i.v. Day 1-3 VP-16 75 mg/m2/d i.v. 1h Day 1-3 cisplatin 75 mg/m2/d i.v. 4h Day 1

   1.1 Courses will be repeated every 28 days for total 2 courses. 1.2 The first and second course will be performed concurrently with radiotherapy.

   1.3 The first course of DEP regimen must be started within one week before or after the initiation of radiation (1st week).

   1.4 The H3-antagonist is permitted for anti-emetic use. 1.5 G-CSF is allowed to be used prophylactically for older ( > 60 years old) patients and for patients with previous or ongoing prolonged myelosuppression.

   Schedule and Dose for DVIP (q4w, post R/T) Dexamethosone 20 mg/m2/d i.v. Day 1-4 VP-16 75 mg/m2/d i.v. 1h Day 1-4 ifosfamide 1.2 mg/m2/d i.v. 2h Day 1-4 mesna 240 mg/m2/d i.v. at 0,4,8 hr Day 1-4 cisplatin 20 mg/m2/d i.v. 1h Day 1-4

   1.6 Courses will be repeated every 28 days for total 2 courses. 1.7 The first course will be performed on the 9th week after the first evaluation of response by CT or MRI.

   1.8 The H3-antagonist is permitted for anti-emetic use. 1.9 G-CSF is allowed to be used prophylactically for older ( > 60 years old) patients and for patients with previous or ongoing prolonged myelosuppression.
2. Involved field radiotherapy Guidelines-

2.1 General Guidelines Local radiation will be given concurrently with chemotherapy from the beginning of treatment. Radiation will be given to the involved field only.

1. Equipment- Only megavoltage equipment with source skin distance of 80 cm, or greater will be used with SAD technique. The treatment cannot be given via electron beam alone even if the lesion is only superficial.
2. Cessation of RT- when any condition of

   1. Grade 4 mucositis with progression.
   2. Grade 4 dermatitis in the RT field with progression
   3. WBC less than 2000/mm3
   4. Infection, which is potentially life threatening.
3. Re-start of RT If toxicity subsides or infection is controlled.

2.2 Target Volume

Gross Tumor Volume (GTV): The GTV is defined as the volume of tumor at presentation as defined by CT, MRI. Uninvolved draining regions are not covered. The treatment cannot be given via electron beam alone even if the lesion is superficial. In cases where there is discrepancy between the scans, the larger volume will be irradiated.

Clinical Target Volume (CTV): This is defined as the GTV with a 1.5cm margin. Include ethmoid sinus and medial half of the maxillary sinus into CTV when gross tumor is located within the nasal cavity. If ethmoid sinus is extensively involved but there is no clinical or radiographic evidence of orbital involvement, the medial bony boundary of the orbit is usually irradiated for possible microscopic disease extension.

Planning Target Volume (PTV): For the purpose of this study, a margin for set up error or patient movement is to be added to the CTV. This may vary but must be at least 0.5cm.

CRITERIA FOR WITHDRAWAL FROM STUDY All patients who are still under or have completed protocol treatments should be continuously followed-up for all study end points. Patients are removed from study if they have completed the protocol or major violations.

1. Completion of assigned therapy and observation.
2. Disease progression.
3. Excessive complication or toxicity.
4. Patient death.
5. Patient withdrawal or refusal.
6. Serum creatinine>3.0 mg/dl
7. Any ≧ grade III toxicity persists ≧ 3 wks after the due day

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven extranodal NK/T-cell lymphoma, nasal type according to the WHO classification (must be pathology-proven EBV DNA positive as well as cytoplasmic CD3 +, while CD56+ is not an essential diagnostic criteria. ). Newly diagnosed patients.
2. Any of lymphomatous involvement exist in nasal cavity and/or paranasal sinuses, orbit, Waldeyer's ring, and oral cavity performance status with ECOG scale 0-2.
3. Stage I or contiguous stage II, measurable or evaluable lymphoma by clinical imaging No previous chemotherapy and/or radiotherapy.
4. ANC ≧ 2,000/mm3, Platelet ≧ 100,000/mm3 of peripheral blood.
5. Age <70.
6. Total bilirubin < 2.5 mg/dl, Serum creatinine ≦1.5 mg/dl, Blood urea nitrogen (BUN) ≦ 25 mg/dl

Exclusion Criteria:

1.Pregnancy or lactation period 2.Severe intercurrent illness, eg. Infection, heart failure 3.Myocardial infarction within recent 12 months 4.Known hypersensitivity to any component drug of the treatment regimen

-

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-05; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
tumor response by CT scan or MRI | the first course of DVIP, one month after the last course of DVIP

SECONDARY OUTCOMES:
EBV DNA level, AEs, Withdrawal from the study treatment | 2-year overall survival and 5-year overall survival , event-free survival, toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Chih Chang, M.D., Principal Investigator — Lymphoma Disease Committee of Taiwan Cooperative Oncology Group
Locations (1):
- National Health Research Institutes, Lymphoma Disease Committee, Taipei, Taiwan

REFERENCES:
- [Derived] Tsai HJ, Lin SF, Chen CC, Chen TY, Su WC, Hwang WL, Lin JC, Chiou TJ, Kao WY, Chiu CF, Chang YF, Chang JS, Chang MC, Su IJ. Long-term results of a phase II trial with frontline concurrent chemoradiotherapy followed by consolidation chemotherapy for localized nasal natural killer/T-cell lymphoma. Eur J Haematol. 2015 Feb;94(2):130-7. doi: 10.1111/ejh.12405. Epub 2014 Oct 10. PMID 24957163